CLINICAL TRIAL: NCT06475534
Title: The Mental Health Experiences of Hispanic and Latinx Dementia Caregivers
Brief Title: The Nuestros Días ("Our Days") Study
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Frank Puga, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: IRB-300008710; 1R01AG072569 (NIH)
Record Dates: First submitted 2024-06-12; First posted 2024-06-26 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Burden; Well-Being, Psychological; Stress, Psychological; Depression; Anxiety
MeSH Terms: conditions — Caregiver Burden; Psychological Well-Being; Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to understand how contextual, individual-level, and cultural factors influence the daily and long-term well-being of caregivers of relatives with memory problems or dementia. The study focuses on caregivers from the Hispanic and Latino community. The main questions it aims to answer are:

* What daily factors increase (i.e., risk factors) or decrease (i.e., protective factors) the daily odds of depression and anxiety symptoms reported by caregivers?
* How do these symptoms vary over time?
* Do variations in depression and anxiety symptoms predict distal health outcomes?

Participants will:

* Complete an online baseline survey to understand their caregiving situation.
* Fill out daily surveys online for three weeks about their caregiving experiences and well-being.
* Complete two follow-up surveys, along with daily surveys, six and twelve months after the baseline survey.

All the study information and surveys can be completed in English or Spanish based on the participant's preference.

DETAILED DESCRIPTION:
Hispanic and Latino/a/x/e (H&L) family caregivers of older relatives living with memory problems or dementia often experience poor mental health due to the increased stress associated with caregiving. The purpose of this study is to examine how contextual, individual-level, and cultural factors influence daily and long-term patterns of depression and anxiety symptoms among H&L caregivers. The investigators will collect data at multiple time points to understand their daily experiences and possible relationships among these factors.

After initial contact, potential participants will complete two eligibility surveys to determine if they are a good fit for the study. If eligible, they will receive a study information sheet outlining all procedures, risks, and benefits.

The study will consist of:

1. Baseline Survey: A 45-minute survey to understand the caregiving situation of each participant.
2. Daily Diaries: After completing the baseline survey, participants will fill out daily surveys for 21 days. These 10-minute surveys will ask about their thoughts, feelings, and experiences of the day and will be emailed at 7 pm each night.
3. Follow-Up Phases: Participants will complete two follow-up phases, one at six months and one at twelve months after the baseline survey. Each phase includes an extended follow-up survey and another series of 21 daily diaries.

The results from this study will inform a dynamic framework of H&L caregiver mental health by identifying modifiable intervention targets associated with resilience over time. This study represents a critical step forward in developing effective, culturally sensitive interventions to support the health and well-being of H&L caregivers, who are often under-supported and face significant challenges in their caregiving role.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Identifies as Hispanic or Latino/a/x/e
3. Provides informal care to a relative living with memory problems or dementia
4. Provides care for 4 hours a day to the person living with memory problems or dementia.

Exclusion Criteria:

1. admission to a nursing home/institutional care for the person living with memory problems or dementia is planned in the next 6 months
2. the potential participant (caregiver) is terminally ill
3. the participant does not have reliable access to the Internet.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of older relatives living with memory problems or dementia who are 18 years or older and Identify as Hispanic or Latino/a/x/e,
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Daily Depression Symptom Experience | 63 days
  Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Depression Short Form, a 4-item scale measuring common symptoms associated with depression.
  Measures common symptoms associated with depression
  4-item Scale 1-5 Likert Scale with 1 indicating "Never" and 5 indicating "Always" Scores range from 4 to 20
  Higher scores indicate higher levels of depressive symptoms
Daily Anxiety Symptom Experience | 63 days
  Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Distress-Anxiety Short Form, a 4-item scale measuring common symptoms associated with anxiety.
  Measures common symptoms associated with anxiety
  4-item Scale 1-5 Likert Scale with 1 indicating "Never" and 5 indicating "Always" Scores range from 4 to 20
  Higher scores indicate higher levels of anxiety symptoms
Depression | 12 months
  Patient Health Questionnaire-9 (PHQ-9), a 9-item scale for screening, diagnosing, monitoring and measuring the severity of depression.
  9-item Scale 0-3 Likert Scale with 0 indicating "Not at all" and 3 indicating nearly every day" Scores range from 0 to 27
  Scores 0 - 4 = Minimal Depression 5 - 9 = Mild Depression 10 - 14 = Moderate Depression 15 - 19 = Moderate Severe Depression 20 - 27 = Severe Depression
Anxiety | 12 months
  General Anxiety Disorder-7 (GAD-7), a 7-item scale for screening, diagnosing, monitoring and measuring the severity of anxiety.
  7-item Scale 0-3 Likert Scale with 0 indicating "Not at all" and 3 indicating nearly every day" Scores range from 0 to 21
  Scores 0 - 4 = Minimal Anxiety 5 - 9 = Mild Anxiety 10 - 14 = Moderate Anxiety >15 = Severe Anxiety
Resilience | 12 months
  Resilience Scale for Adults: a 33-item scale measuring personal competence, social competence, personal structure, family coherence, and social support.
  14-item scale with 3 subscales (Perception of self, planned future, structured style) 1-7 Likert Scale with 1 indicating "Not true at all" and 7 indicating "Very true"
  Higher scores indicate higher levels of resilience in the indicated subcategory
Health Related Quality of Life | 12 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health: 10 item scale measuring global health-related quality of life (HRQOL) across 2 domains: physical and mental health.
  10-item Scale 9 Items use 0 to 4 Likert Scale Item 10: 0 to 10 Likert Scale that is recoded to five categories (0 = 1; 1-3 = 2; 4-6 = 3; 7-9 = 4; 10 = 5) Scores range from 0 to 41
  Higher scores indicate better overall mental and physical health

CONTACTS AND LOCATIONS:
Overall Officials: Frank Puga, PhD, Principal Investigator — Univeristy of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No